CLINICAL TRIAL: NCT01119521
Title: Phase I Study of Whether Preclearance of Latent M. Tuberculosis (MTB) Infection With Isoniazid (INH) Enhances Specific Immune Responses to MTB Following Subsequent BCG Revaccination in Healthy, HIV-Uninfected, Tuberculin Skin Test Positive Adults
Brief Title: Study of Pre-clearance of Latent Tuberculosis Infection And BCG Revaccination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07-0083
Record Dates: First submitted 2010-04-29; First posted 2010-05-07 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-12

CONDITIONS: Tuberculosis
Keywords: South Africa,tuberculosis,vaccine
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid

ARMS (2):
- Group A: INH; BCG (Experimental): 6 months of Isoniazid (INH) treatment for latent tuberculosis infection (LTBI) (completed within no more than 7 months) followed by intradermal Bacillus Calmette-Guérin (BCG) revaccination.
  Interventions: Biological: BCG strain Danish; Drug: Isoniazid
- Group B: observation; BCG; observation; INH (Experimental): 7 months of observation (run in period) followed by intradermal Bacillus Calmette-Guérin (BCG) revaccination followed after 6 months of observation by 6 months of Isoniazid (INH) treatment for latent tuberculosis infection (LTBI).
  Interventions: Biological: BCG strain Danish; Drug: Isoniazid

INTERVENTIONS:
Biological: BCG strain Danish — Intradermal Bacillus Calmette-Guerin (BCG) live-attenuated vaccine prepared using the Danish 1331 BCG substrain; adult dose contains 2 to 8 x 10^5 colony forming units (CFU) BCG.
Drug: Isoniazid — United States Pharmacopeia 100 mg or 300 mg oral tablets [5 mg/kilogram/day (rounded up to nearest 100 mg; maximum dose 300 mg/day)].

SUMMARY:
The purpose of this research is to further study the tuberculosis (TB) vaccine, Bacillus Calmette Guérin (BCG). The goal of this study is to evaluate whether the BCG vaccine is more effective in preventing TB in adults if it is given after 6 months of treatment with a widely used anti-TB drug, isoniazid (INH). Participants will include 82 healthy, tuberculin skin test positive (TST+), HIV-uninfected, male and female volunteers, aged 18-40 years. The study will be conducted in Worcester, South Africa. Subjects will be assigned by chance to 1 of 2 possible treatment groups. Group 1 will receive 6 months of oral INH treatment followed by intradermal (administered into the skin) BCG revaccination and one year of follow-up. Group 2 will be observed for 7 months which will be followed by intradermal BCG revaccination and another 6 months of follow-up. Then 6 months of INH treatment will be given. Participants will be involved in study procedures for about to 22 months.

DETAILED DESCRIPTION:
This study is a phase I, single-center, open label, randomized controlled clinical trial assessing the effect of pre-clearance of latent Mycobacterium tuberculosis (MTB) by Isoniazid, isonicotinic acid hydrazine (INH) treatment before Bacillus Calmette-Guérin (BCG) revaccination versus BCG revaccination alone on mycobacterial-specific immune responses in tuberculin skin test (TST) positive adults. Subjects initially assigned to observation prior to BCG revaccination will receive INH treatment of latent tuberculosis infection (LTBI) beginning six months after revaccination. Volunteers will include 82 healthy, TST positive human immunodeficiency virus (HIV)-uninfected, male and female persons aged 18-40 years. The primary objectives of the study are to: determine the effect of INH preclearance on the kinetics and characteristics of the specific immune response following BCG revaccination in adults with latent MTB infection (TST positive); and determine the safety and reactogenicity of BCG revaccination in TST positive adults. The secondary objectives of the study are to: determine the effect of INH preclearance and BCG revaccination on MTB-specific Th1 effector and central memory cell function; determine the effect of INH preclearance and BCG revaccination on MTB-specific Treg cell function; and determine the effect of INH preclearance and BCG revaccination on innate immune responses as measured by T cell mediated inhibition of intracellular mycobacterial growth and inflammatory cytokine production. All subjects are expected to be enrolled over 12 months. The duration of screening, enrollment, and follow-up for subjects is up to 22 months. Subjects will be randomly assigned to receive either: 6 months of INH treatment for LTBI (completed within no more than 7 months) followed by intradermal BCG revaccination or 7 months of observation (run in period) followed by intradermal BCG revaccination followed after 6 months of observation by 6 months of INH treatment for LTBI. Both groups will receive their BCG vaccinations during the same time period. Volunteers will be evaluated at 7 and 14 days and 1, 3, 6 and/or 12 months after BCG revaccination and each month of INH therapy and the end of study for safety, reactogenicity and immunogenicity. Blood for immunologic studies will be drawn at study enrollment for subjects, just prior to BCG revaccination, and 1, 2 weeks and 1, 3 and either 6 or 12 months (depending on which study arm) after BCG vaccination, and months 1, 3, 6 of INH therapy and the end of study for measurement of MTB specific T cell responses. Both treatment arms will be followed for safety and immunogenicity endpoints for 12 months after BCG revaccination. Immunologic outcomes have been chosen with the goal of measuring the characteristics and kinetics of human immune responses following BCG vaccination to support the ultimate aim of developing methods to determine the biological relevance of immune responses induced by BCG revaccination and their relevance to protection from tuberculosis (TB). Overall, this study may provide key information on the characteristics and kinetics of immune responses following BCG revaccination in adults and whether these are affected by preclearance with INH treatment of LTBI.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant, non-lactating females aged 18 to 40 years, inclusive.
2. Be available for study follow-up.
3. Be in good general health as judged by a physician on the basis of reported medical history and physical examination including blood pressure (BP) and respiratory evaluation.
4. Have a visible Bacillus Calmette-Guérin (BCG) scar. Subjects with medical documentation of BCG vaccination after 2 years of age will be excluded.
5. Have a positive (greater than or equal to 15 mm induration at 48 to 72 hours after placement) tuberculin skin test [TST; Mantoux method using 2 tuberculin units (TU) Purified Protein Derivative (PPD) RT-23].
6. Weigh at least 45 kg.
7. Negative human immunodeficiency virus (HIV) approved test.
8. Demonstrate adequate understanding of the study and its requirements for participation, as demonstrated by discussions with study staff, and be able to provide written informed consent to participate in the study.
9. Females must not be pregnant, as determined by negative pregnancy test at screening, have a negative urine pregnancy test on the day of BCG revaccination, and must be non-lactating. For women of child bearing potential, use an effective contraception (licensed hormonal treatment, monogamous relationship with vasectomized partner, surgical sterilization) for 30 days prior to immunization and for the 2-year period of study follow-up.
10. Serum aspartate aminotransferase (AST) or alanine transaminase (ALT) < 1.1 x upper limit of normal (ULN) and serum total bilirubin < 1.1 x ULN.
11. Serum creatinine < 1.5 mg/dL; urinalysis dipstick negative for glucose and 1 plus protein.
12. Total white blood cell (WBC) count > 3.5 x 10^3/mm^3 and < 10.8 x 10^3/mm^3.
13. Hemoglobin > 12 gm/dL (female) and > 13.5 gm/dL (male).
14. Have negative serologic tests for hepatitis B surface antigen and hepatitis C antibody.

Exclusion Criteria:

1. Known hypersensitivity to Isoniazid (INH) or to any component of Bacillus Calmette-Guérin (BCG) vaccine.
2. Exposure to a case of Tuberculosis (TB) with known INH resistance.
3. Current smear or culture-confirmed or clinically diagnosed active TB
4. Suspected active TB (recurrent fever, fatigue, night sweats, weight loss, oral ulcers, diarrhea, nausea or vomiting, bleeding) or patients who are receiving anti-tuberculosis drugs.
5. Prior TB treatment, prior treatment for latent tuberculosis infection (LTBI), a self-reported history or vaccination card or medical record documenting receipt of BCG vaccination after 2 years of age.
6. Pregnant or nursing females.
7. Chronic immunosuppressive disorder or a condition requiring chronic immunosuppressive treatment such as rheumatoid arthritis or severe asthma requiring chronic corticosteroid therapy. For corticosteroids, this will mean prednisone, or equivalent, 0.5 mg/kg/day or daily use of inhaled corticosteroids. Topical steroids are allowed.
8. Active dermatitis such as atopic dermatitis.
9. Persons with any history of scarring badly or keloid formation based on physical examination.
10. Receipt of blood products or immunoglobulin within six months of BCG revaccination.
11. History of chronic illness requiring close physician follow up, including known chronic liver disease or cirrhosis, or any medical, psychiatric, occupational, or substance abuse problems that make it unlikely the volunteer will comply with the protocol as determined by the local investigator.
12. History of acute or chronic medical conditions including, but not limited to diabetes mellitus, chronic renal failure/dialysis, silicosis, gastrectomy, jejunoileal bypass, solid organ transplantation such as renal or cardiac transplants, carcinoma of the head and neck, and disorders of the liver, kidney, lung, heart, or nervous system, or other metabolic or autoimmune/inflammatory conditions.
13. Have any systemic symptoms including fever, myalgia, fatigue, chills, night sweats, weight loss, nausea, vomiting or bleeding, diarrhea, abdominal pain, rhinorrhea, cough, wheezing, or shortness of breath within 72 hours before vaccination or signs of mucosal ulceration, lymphadenitis, gastrointestinal, or pulmonary disease by physical examination on day of vaccination. Subjects with minor self-limited illnesses such as common colds or gastroenteritis may return for re-evaluation after 3 days if their symptoms have abated for vaccination.
14. Have lymphadenopathy, hepatosplenomegaly, or other abnormalities on physical examination.
15. Have close contacts, with confirmed or suspected, human immunodeficiency virus (HIV) infection or other immunodeficiency state (including diabetes mellitus, chronic dermatitis/severe eczema, chronic renal failure, hematologic malignancy), or on chronic immunosuppressive therapy. A close contact is defined as a person who lives in the same home as the subject.
16. Live in a household where any household member has been diagnosed or treated for active TB during the previous 2 years.
17. Have received or currently be receiving chronic (more than 14 days) immunosuppressive therapy within 6 months prior to screening. This includes chronic treatment with oral prednisone 0.5 mg/kg/day (or equivalent). Inhaled and topical steroids are allowed.
18. Persons with chronic heavy ethanol intake or injection drug use. Chronic heavy ethanol intake is defined as an average continuous daily intake of more than 2 drinks, or a pattern of ethanol use, which, in the opinion of the investigator would prejudice his or her participation in the trial. Injection drug use will be defined as any non-medical injection drug use during the previous 2 years.
19. Participated in another research study that includes receiving an experimental drug within 30 days prior to study entry.
20. Receipt of live attenuated vaccines within 60 days of study entry. Note: Medically indicated inactivated vaccines are not exclusionary, but should be given at least 2 weeks away from BCG revaccination, or any immunologic sampling time point post BCG revaccination.
21. Have a history of the use of a systemic antibiotic within the 14 days prior to revaccination or planned use of a systemic antibiotic in the 3 months after revaccination.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2010-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Adverse reactions/events [and whether they meet the definition of a serious adverse event (SAE)], the severity of these reactions, and related measurements, and assessed relationship to vaccine administration. | 1, 3, 7 and 14 days and 1, 3, 6 and/or 12 months after BCG revaccination and each month of INH therapy, up to 22 months.
Direct Ex-vivo gene expression signature (RNA) | At baseline, day 1, 3, and week 1 following BCG vaccination
Effector T cell function by whole blood cytokine production (WBA),flow cytometric measures of intra-cellular cytokine production (ICS) or ELISA assays to measure immune function | Enrollment, baseline, Week 1 and 2, Months 1, 3 and 6 after BCG vaccination, and Month 1, 3 and 6 of INH therapy.
Memory T cell function by whole blood cytokine production (WBA),flow cytometric measures of intra-cellular cytokine production (ICS) or ELISA assays to measure immune function. | Enrollment, baseline, Week 1 and 2, Months 1, 3 and 6 after BCG vaccination, and Month 1, 3 and 6 of INH therapy.
Precursor frequencies of mycobacterial antigen-specific T cells will be measured by ELISPOT using standard methods and SOPs | Enrollment, baseline, Week 1 and 2, Months 1, 3 and 6 after BCG vaccination, and Month 1, 3 and 6 of INH therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cape Town - Institute of Infectious Disease and Molecular Medicine, Cape Town, Western Cape, South Africa

REFERENCES:
- [Result] Suliman S, Geldenhuys H, Johnson JL, Hughes JE, Smit E, Murphy M, Toefy A, Lerumo L, Hopley C, Pienaar B, Chheng P, Nemes E, Hoft DF, Hanekom WA, Boom WH, Hatherill M, Scriba TJ. Bacillus Calmette-Guerin (BCG) Revaccination of Adults with Latent Mycobacterium tuberculosis Infection Induces Long-Lived BCG-Reactive NK Cell Responses. J Immunol. 2016 Aug 15;197(4):1100-1110. doi: 10.4049/jimmunol.1501996. Epub 2016 Jul 13. PMID 27412415
- [Result] Johnson JL, Geldenhuys H, Thiel BA, Toefy A, Suliman S, Pienaar B, Chheng P, Scriba T, Boom WH, Hanekom W, Hatherill M. Effect of isoniazid therapy for latent TB infection on QuantiFERON-TB gold in-tube responses in adults with positive tuberculin skin test results in a high TB incidence area: a controlled study. Chest. 2014 Mar 1;145(3):612-7. doi: 10.1378/chest.13-1232. PMID 24135768
- [Result] Hatherill M, Geldenhuys H, Pienaar B, Suliman S, Chheng P, Debanne SM, Hoft DF, Boom WH, Hanekom WA, Johnson JL. Safety and reactogenicity of BCG revaccination with isoniazid pretreatment in TST positive adults. Vaccine. 2014 Jun 30;32(31):3982-8. doi: 10.1016/j.vaccine.2014.04.084. Epub 2014 May 9. PMID 24814553
- [Derived] Suliman S, Murphy M, Musvosvi M, Gela A, Meermeier EW, Geldenhuys H, Hopley C, Toefy A, Bilek N, Veldsman A, Hanekom WA, Johnson JL, Boom WH, Obermoser G, Huang H, Hatherill M, Lewinsohn DM, Nemes E, Scriba TJ. MR1-Independent Activation of Human Mucosal-Associated Invariant T Cells by Mycobacteria. J Immunol. 2019 Dec 1;203(11):2917-2927. doi: 10.4049/jimmunol.1900674. Epub 2019 Oct 14. PMID 31611259
- [Derived] Scriba TJ, Penn-Nicholson A, Shankar S, Hraha T, Thompson EG, Sterling D, Nemes E, Darboe F, Suliman S, Amon LM, Mahomed H, Erasmus M, Whatney W, Johnson JL, Boom WH, Hatherill M, Valvo J, De Groote MA, Ochsner UA, Aderem A, Hanekom WA, Zak DE; other members of the ACS cohort study team. Sequential inflammatory processes define human progression from M. tuberculosis infection to tuberculosis disease. PLoS Pathog. 2017 Nov 16;13(11):e1006687. doi: 10.1371/journal.ppat.1006687. eCollection 2017 Nov. PMID 29145483